CLINICAL TRIAL: NCT01187069
Title: A Practice-nurse Addressed Intervention to Improve Type 2 Diabetes Care. A Pragmatic Cluster Randomised Controlled Trial in Primary Health Care
Brief Title: A Practice-nurse Addressed Intervention to Improve Type 2 Diabetes Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: TrygFonden, Denmark (Industry); Sygekassernes Helsefond (Other); Lundbeck Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2009-41-3065
Record Dates: First submitted 2010-06-14; First posted 2010-08-23 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Type 2 Diabetes
Keywords: Motivation; patients with type 2 diabetes; practice nurses; general practice; Self-determination Theory
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Training course for practice nurses in autonomy support (Experimental)
  Interventions: Behavioral: Training course for practice nurses in autonomy support
- Control (No Intervention): Control practices were randomly drawn from among intervention practice applicants and were informed by mail about their status as control practice.

INTERVENTIONS:
Behavioral: Training course for practice nurses in autonomy support — An interactive course consisting of 4X4 hours education in autonomy support over a 6 months period. The main-components in the course are 1) communication skills, 2) introduction to patient work-sheets and 3) a quick up-to-date knowledge about treatment recommendations of type 2 diabetes. Furthermore, the nurses in the intervention-practices receive a half an hour support-visit 4-5 months after the end of the course.
  Arms: Training course for practice nurses in autonomy support

SUMMARY:
A huge challenge in type 2-diabetes care is how to motivate patients towards health behaviour changes. In Denmark, the tendency is that nurses in general practice provide a large part of type 2 diabetes care.

Observational studies support Self-determination Theory by finding autonomous motivation and perceived competence associated with improved HbA1c-levels in patients with type 2 diabetes. Hence, research is needed to develop and test interventions that are autonomy supportive.

Aim To develop a training course for practice-nurses in autonomy support in patients with type 2 diabetes, and to evaluate the effect on patient outcomes.

Methods The development of the intervention was based on literature research and expert meetings. The intervention is evaluated in a cluster randomised controlled trial with 40 Danish general practices,

* where nurses, before enrolment in the study, provided consultations to patients with type 2 diabetes,
* and about 2500 patients with type 2 diabetes, identified in a Diabetes Database.

The patients will be followed 15 months from nurse-participation in the course. Data will be obtained from registers and patient-questionnaires. The hypothesis is that patients with type 2 diabetes regardless of education level, age, and gender will benefit from the intervention.

ELIGIBILITY:
Inclusion Criteria:

* The intervention-study comprises 40 general practices were:

  1. more than 50% of the patients with type 2 diabetes, who had participated in diabetes-consultations during the last year from the invitation-date to the project, were seen by a nurse at least once, stated by the practice. The diabetes-consultation should not only include examinations (blood tests and blood pressure measurement), but should also include communication about living with type 2 diabetes ;
  2. enrollment in the project before registration deadline (three weeks after invitation).

Patients with diabetes, alive and affiliated the practices by May 2011, were identified in a a validated diabetes database based on health registers; The national Patient Registry, The national Health Insurance Service registry, the prescription database and the laboratory database in the county.

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
HbA1c | Last measurement within 12 months before - and 15 months after nurse participation in the course
  Collected from registers (historical data - not measured as a part of this study)

SECONDARY OUTCOMES:
HDL-cholesterol | Last measurement within 12 months before - and 15 months after nurse participation in the course
  Collected from registers (historical data - not measured as a part of this study)
LDL-cholesterol | Last measurement within 12 months before - and 15 months after nurse participation in the course
  Collected from registers (historical data - not measured as a part of this study)
Perceived autonomy support (HCCQ) | 15 months from nurse participation in the course
  Modified health care climate quastionaire (Self-determination Theory)
Type of motivation (TSRQ) | 15 months from nurse participation in the course
  The treatment self-regulation quastionaire (Self-determination Theory)
Perceived competence (PCS) | 15 months from nurse participation in the course
  perceived competence scale (Self-determination Theory)
Total-cholesterol | Last measurement within 12 months before - and 15 months after nurse participation in the course
  Collected from registers (historical data - not measured as a part of this study)
Self-rated health (SF-12) | 15 months from nurse participation in the course
Problem Areas In Diabetes scale (PAID) | 15 months from nurse participation in the course

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Practice, School of Public Health, Aarhus University, Aarhus, Denmark

REFERENCES:
- [Derived] Juul L, Maindal HT, Zoffmann V, Frydenberg M, Sandbaek A. Effectiveness of a training course for general practice nurses in motivation support in type 2 diabetes care: a cluster-randomised trial. PLoS One. 2014 May 5;9(5):e96683. doi: 10.1371/journal.pone.0096683. eCollection 2014. PMID 24798419
- [Derived] Juul L, Maindal HT, Zoffmann V, Frydenberg M, Sandbaek A. A cluster randomised pragmatic trial applying Self-determination theory to type 2 diabetes care in general practice. BMC Fam Pract. 2011 Nov 24;12:130. doi: 10.1186/1471-2296-12-130. PMID 22111524